CLINICAL TRIAL: NCT06857305
Title: Efficacy and Safety of Biweekly Regimen of Eribulin Versus a Standard Regimen for the Treatment of Locally Recurrent or Metastatic HER2-negative Breast Cancer: a Multicenter, Randomized, Open-label, Phase III Trial
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ma Fei，MD (Other)
Responsible Party: Sponsor-Investigator, Ma Fei，MD, Cancer Hospital Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4143
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eribulin biweekly regimen (Experimental)
  Interventions: Drug: Eribulin biweekly regimen
- eribulin standard regimen (Experimental)
  Interventions: Drug: Eribulin standard regimen

INTERVENTIONS:
Drug: Eribulin biweekly regimen — Eribulin biweekly regimen
  Arms: eribulin biweekly regimen
Drug: Eribulin standard regimen — Eribulin standard regimen
  Arms: eribulin standard regimen

SUMMARY:
Eribulin is a soft spongin-like inhibitor of mitotic microtubule dynamics in cells. From the evidence of efficacy, the STUDY 305 and STUDY 301 studies suggest that eribulin improves PFS and OS in patients with breast cancer. Eribulin has a good safety profile with a low incidence of patient-perceivable adverse effects, with myelosuppression being the main adverse effect, and neutropenia, anemia, and also fatigue being the most common adverse effects. However, serious neutropenia, may result in delayed dosing, dose reduction or discontinuation in some patients.

In studies of standard regimen therapy with eribulin, grade 3-4 neutropenia occurred in approximately 45% of patients, of which approximately 25% required dose adjustment or discontinuation of therapy, which has become an urgent clinical problem in the treatment of eribulin. Therefore, a modified bi-weekly regimen of eribulin (1.4 mg/m2 intravenously on days 1 and 15 of a 28-day cycle), based on the standard regimen (1.4 mg/m2 intravenously on days 1 and 8 of a 21-day cycle), is expected to improve the safety of eribulin administration without compromising efficacy, in order to minimize dose reductions of the medication and interruptions of therapy, thereby improving patients' quality of life.

There is still a lack of head-to-head studies on the efficacy and safety of the combination of eribulin standard regimen and biweekly regimen in HER2-negative advanced breast cancer, and the treatment data in the Chinese population need to be further explored. The aim of this study is to explore the efficacy and safety of eribulin biweekly regimen compared with the standard regimen in patients with locally recurrent or metastatic HER2-negative breast cancer, and to provide a clinical evidence-based basis for the optimization of eribulin treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. ECOG 0-2
3. Expected survival of not less than 12 weeks
4. At least one measurable lesion
5. With HER2 negative locally recurrent or metastatic breast cancer
6. Metastatic breast cancer advanced stage received ≤3 lines of chemotherapy
7. Previous anthracycline and paclitaxel therapy
8. Well organ functional status 1）routine blood test

   * ANC≥1.5×109/L；
   * PLT≥90×109/L；
   * Hb≥90 g/L； 2）blood biochemistry
   * TBIL≤1.5×ULN；
   * ALT/AST≤2×ULN；patients with liver matastasis ALT/AST≤5×ULN；
   * BUN/Cr≤1.5×ULN and creatinine clearance ≥50 mL/min （Cockcroft-Gault） 3）cardiology ultrasound
   * LVEF≥50%；
9. Signed informed consent, good compliance and willingness to cooperate with follow-up visits

Exclusion Criteria:

1. With third interstitial fluid that cannot be controlled by drainage or other means
2. Symptomatic brain or meningeal metastases
3. Patients with only bone or skin as the sole target lesion
4. Pre-existing other malignant tumors
5. Patients who have used eribulin in the adjuvant and palliative phases of care
6. Known history of allergy to components of this regimen; history of immunodeficiency
7. Pregnant or breastfeeding female patients, female patients of childbearing potential with a positive baseline pregnancy test or female patients of childbearing potential who are unwilling to use effective contraception throughout the trial period
8. Have a concomitant illness that, in the investigator's judgment, seriously jeopardizes the patient's safety, or interferes with the patient's ability to complete the study.
9. A clear past history of neurological or psychiatric disorders
10. Any other condition for which the investigator believes the patient is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate | From enrollment to the end of treatment at 8 weeks
  Clinical benefit was defined as patients who achieve complete response/partial response or stable disease of over 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongnan Mo, Study Chair — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Hospital Chinses Academy of Medical Sciences, Beijing, B, China